CLINICAL TRIAL: NCT00242827
Title: An Open-Label Study of the Efficacy and Safety of Oral CEP-701 for the Treatment of Patients With Advanced Multiple Myeloma
Brief Title: Efficacy and Safety of Oral CEP-701 for the Treatment of Patients With Advanced Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C0701/2025/ON/US
Record Dates: First submitted 2005-09-27; First posted 2005-10-21 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2006-09

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — lestaurtinib

INTERVENTIONS:
Drug: Oral CEP-701

SUMMARY:
An Open-Label Study of the Efficacy and Safety of Oral CEP-701 for the Treatment of Patients with Advanced Multiple Myeloma.

DETAILED DESCRIPTION:
An Open-Label Study of the Efficacy and Safety of Oral CEP-701 for the Treatment of Patients with Advanced Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if all of the following criteria are met:

* Histological and cytological confirmation of stage II or III multiple myeloma.
* Relapsed or primary refractory multiple myeloma, after 1 or more courses of standard therapy, and progressive disease.
* ECOG performance status of 0-1.
* Measurable disease as defined by serum M protein of more than 1.0 gm/dl, serum light chain of more than 200 mg/dL, or Bence-Jones proteinuria of more than 200mg/24 hours.
* At least 18 years of age.
* Normal marrow function: ANC>1.0x10 9/L, platelets>50X10 9/L An exception is allowed if myelosuppression or thrombocytopenia is secondary to bone marrow plasmacytosis. Growth factor support is allowed.
* Normal organ function: bilirubin <1.5XULN, AST and ALT<2XULN, serum creatinine <2.0 mg/dL.
* Contraceptive measures during participation as appropriate.
* Willing to be able to comply with study procedures and restrictions.
* Signed written informed consent.

Exclusion Criteria:

Patients are excluded from participating in this study if 1 or more of the following criteria are met:

* Nonsecretory disease or plasma cell leukemia (defined as >2000 circulating plasma cells/uL).
* More than 4 prior courses if anticancer therapy (bisphosphonates are not considered anticancer therapy for this criterion)
* Chemotherapy or radiotherapy within 4 weeks prior to enrollment
* Unresolved adverse events or uncontrolled illness that would be likely to interfere with the objectives of the study.
* Treatment with an investigational drug within 4 weeks of first day of study treatment
* History of second cancer (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free more than 5 years).
* Treatment with potent CYP3A4 inhibitors including cyclosporine, clotrimazole, fluconazole, itraconazole, ketoconazole, voriconazole, erythromycin, clarithromycin, and troleandomycin, human immunodeficiency virus (HIV), protease inhibitors, or nefazodone within 1 week (7 days) of the planned 1st day of study treatment.
* Currently receiving warfarin.
* Clinical diagnosis of active gastrointestinal ulceration of melena or hematemesis in the previous 4 weeks.
* Hypersensitivity to CEP701 or any component of CEP701.
* Intolerance of dexamethasone.
* Requirement for HIV protease inhibitor treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-04; Study Completion 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brown, Study Director — Cephalon
Locations (5):
- United States (5):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Indiana Univeristy Cancer Research Center, Indianapolis, Indiana
  - The Cancer Center Hackensack University Medical Center, Hackensack, New Jersey
  - New York Presbyterian Hospital, New York, New York
  - Abramson Cancer Center Of University of Pennsylvania, Philadelphia, Pennsylvania